CLINICAL TRIAL: NCT05921097
Title: Comparison of Histamine and Local Heating for Evoking the Axon-reflex Flare Response in Diabetes
Acronym: HistaHeat
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Johan Bovbjerg Røikjer, Postdoc, Aalborg University Hospital
Other Study IDs: N-20230007
Record Dates: First submitted 2023-06-07; First posted 2023-06-27 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetic Neuropathy Peripheral; Small Fiber Neuropathy
Keywords: Diabetes; Neuropahty
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Small Fiber Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T1DM: People with type 1 diabetes
  Interventions: Diagnostic Test: Histamin-induced axon-reflex flare response; Diagnostic Test: Local heating-induced axon-reflex flare response; Diagnostic Test: 2-point discrimination tasks; Diagnostic Test: NC-Stat DPNCheck; Diagnostic Test: QST; Diagnostic Test: Biothesiometry

INTERVENTIONS:
Diagnostic Test: Histamin-induced axon-reflex flare response — Histamin-induced axon-reflex flare response
Diagnostic Test: Local heating-induced axon-reflex flare response — Local heating-induced axon-reflex flare response
Diagnostic Test: 2-point discrimination tasks — 2-point discrimination tasks
Diagnostic Test: NC-Stat DPNCheck — NC-Stat DPNCheck
Diagnostic Test: QST — QST
  Other Names: Quantitative Sensory Testing, thermal
Diagnostic Test: Biothesiometry — Biothesiometry
  Other Names: VPT

SUMMARY:
Diabetic peripheral neuropathy is the most common complication to diabetes mellitus affecting as much as 50% of the population with diabetes. Symmetrical sensory neuropathy is by far the most common pattern, which often progress slowly over many years, although some individuals experience faster and more severe courses. Despite the frequent occurrence, the causes of diabetic peripheral neuropathy are largely unknown, which is reflected in the fact that no disease-modifying treatments are available for preventing, treating or even halting the progression of the disease. The consequences can be dire, as neuropathy frequently leads to foot ulcers, amputations or intolerable neuropathic pain in the lower extremities. Sensory loss may go completely undetected in diabetes, as there often are literally no symptoms. For many individuals, the development of diabetic peripheral neuropathy can therefore proceed completely unnoticed, making regular screening the most important tool for diagnosing the condition. Unfortunately, unlike nephropathy or retinopathy, diabetic peripheral neuropathy is not easily screened for, as the condition lacks reliable markers for early- or progressing disease. Therefore, screening for diabetic peripheral neuropathy currently revolves around diagnosing loss of protective sensation, judged by the inability to feel vibration or light touch. However, in their most recent guidelines, the American Diabetes Association has included screening for small fibre neuropathy using either the cold- and heat perception thresholds or pinprick as a clinical standard. Although this acknowledgement of the importance of assessing not only large- but also small nerve fibres is a huge step towards early detection of diabetic peripheral neuropathy, the overriding issue of insensitive, unreproducible, and inaccurate bedside tests for small nerve fibres remains. While cold- and heat perception and pinprick sensation are indeed mediated by small nerve fibres, the sensitivity of these methods, outside of extreme standardization only achievable in dedicated neuropathy research-centres, remain poor and not usable on an individual level. This lack of sensitivity has also become apparent in several large clinical trials, where the methods have continuously failed as robust clinical endpoints. Due to this, the hunt for a sensitive and reproducible method for adequate assessment of the small nerve fibres have begun. Amongst several interesting methods, two have gained particular interest (corneal confocal microscopy and skin biopsies with quantification of intra-epidermal nerve fiber density), due to their diverse strengths, although clinical application is currently limited to a few specialized sites. Furthermore, both methods suffer several inherent issues including that fact that they only provide information about the structure of the nerves and not the function. One method to assess the function of small cutaneous C-fibers is the assessment of the axon reflex flare response using laser doppler imaging (LDI) or Full-field laser perfusion imaging (FLPI), which has classically been studied using local heating. Unfortunately, this method is limited in clinical usage due to time-consumption. The investigators recently published an alternative method using a simple skin-prick application of histamine to evoke the response, which reduced the examination-time markedly. Before claiming the method to be a better alternative, the investigators do however need to prove that the method is as good as the original.

In addition to the direct comparison of the histamine-induced and the heating-induced axon-reflex flare response the study will also assess spatial acuity in the same cohort as a secondary aim. Spatial acuity is considered as a measure of the sensory systems ability to code spatial information regarding an external stimulus. To investigate the spatial acuity, the 2-point discrimination task (2PDT) is often used. Spatial acuity has been shown to be impaired in several chronic pain condition. Additionally, it has been shown that the 2PDT may be a useful tool to understand the sensory changes in diabetes[8].

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years and diagnosed with type 1 diabetes

Exclusion Criteria:

* Known critical limb ischemia (ankle-brachial index < 50 mmHg or toe-brachial index < 30 mmHg)
* Symptoms of claudicatio intermittens
* Inability to do without antihistamine for 24h prior to examination
* Known neurological disease (e.g., multiple sclerosis)
* Severe skin diseases on either foot (e.g., fulminant pemphigoid)
* Previous or current alcohol or drug abuse
* Previous or current chemotherapy or current disseminated cancer
* Known cause of neuropathy other than diabetes
* Previous amputation on either foot
* Active diabetic foot ulcer on either foot
* Pregnancy
* Inability to participate or other condition thought to impact the results (evaluated by investigator)
* Asymmetrical neuropathy (i.e., previous accident with radiating pain)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with T1DM
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-06-17 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Comparison of histamine and local heating (area size) | Through study completion, an average of 1-2 years
  The evoked area (assessed by full-field laser speckle perfusion imaging) by histamine and local heating will be compared as a proxy for small fiber neuropathy in diabetes
Comparison of axon-reflex flare responses with QST | Through study completion, an average of 1-2 years
  Comparison of axon reflex flare responses with an established method (area size vs cold and heat detection threshold)

SECONDARY OUTCOMES:
2PDT in diabetes with and without DPN | Through study completion, an average of 1-2 years
  Assess spatial acuity through 2PDT in people with diabetes with and without DPN.
Comparison of axon-reflex flare responses with NC-Stat DPNCheck | Through study completion, an average of 1-2 years
  Comparison of axon reflex flare responses with an established method (sural nerve conduction velocity/amplitude)

OTHER OUTCOMES:
Exploratory | Through study completion, an average of 1-2 years
  This endpoint will report correlations between the different methods used in the study. These correlations are exploratory and not predetermined
DPN severity and pain | Through study completion, an average of 1-2 years
  Correlations between DPN severity (including pain) and methods

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No